CLINICAL TRIAL: NCT05394571
Title: Conditions Associated With Poorly Controlled Diabetes in Patients With Type 2 Diabetes and Early Changes in HbA1c Values With Tailored Treatment
Brief Title: Conditions Associated With Poorly Controlled Diabetes in Patients With Type 2 Diabetes and HbA1c Changes With Therapy
Status: Completed | Type: Observational
Sponsor: Goztepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayse N Erbakan, Principal Investigator, Goztepe Training and Research Hospital
Other Study IDs: Poorly controlled T2DM
Record Dates: First submitted 2022-05-19; First posted 2022-05-27 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Type 2 Diabetes; Poorly Controlled Diabetes Mellitus
Keywords: type 2 diabetes; poorly controlled Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Newly diagnosed diabetes: Patients who have been diagnosed with type 2 diabetes within a month
- Had controlled diabetes before: Patients who had at least two HbA1c levels =<%7,5 before enrollment
- Had moderately uncontrolled diabetes: Patients who had at least two HbA1c levels between %7,5 and %9,49 before enrollment
- Had poorly controlled diabetes: Patients who had at least two HbA1c levels above %9,5 before enrollment

SUMMARY:
In Turkey, only 55% of patients with type 2 diabetes have been diagnosed, and 91% of these patients have been receiving treatment. The rate of patients reaching the treatment target is 50%. The pandemic has also affected diabetic patients. We aimed to determine the characteristics of patients with type 2 diabetes (HbA1c >=10) with poor metabolic control and to evaluate the extent to which metabolic control can be achieved in 3 months.

DETAILED DESCRIPTION:
Patients who applied to Istanbul Medeniyet University Goztepe Prof. Dr. Suleyman Yalcin City Hospital Diabetes Polyclinics and have an HbA1c levels of >= 10% in their examinations will be admitted to the study. Detailed history, including medication usage and previous blood tests will be questioned. The patients will be asked to complete questionnaires about their eating patterns (mindful eating questionnaire), their physical activities (General practice physical activity questionnaire), and whether they have depression (Beck depression questionnaire).

Anthropometric measurements will be taken, and biochemical data will be recorded. Patients will be grouped according to their previous HbA1c values as a) newly diagnosed, b) those whose diabetes was previously controlled, c) those whose diabetes was previously not at the target range but now worsened, and d) those whose diabetes was poorly controlled from the beginning.

Diabetes follow-up will be continued by their respective physicians. The patients will be called again three months after their enrollment to record the most recent biochemical data. Patient characteristics (age, gender, educational status, depression status, eating awareness, exercise characteristics) will be evaluated in accordance with the predetermined HbA1c groups. Again, according to the patient groups, the difference in HbA1c after three months, the frequency of reaching the target, and possible factors associated with the findings will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 2 diabetes
* give consent to the study
* accessibility to the previous and recent test results

Exclusion Criteria:

* acute infection or inflammation lasting more than a week
* acute metabolic decompensation
* unable to attend to the follow-ups
* having non-thyroid endocrine diseases
* active oncologic treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with type 2 diabetes and have an HbA1c level equal to or higher than 10%
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in HbA1c levels after 3 months treatment | Three months
  Changes in HbA1c levels after 3 months treatment according to the predetermined HbA1c groups.
Changes in HbA1c levels equal to or more than 20% | Three months
  Comparison of the patient groups according to the reduction of 20% or more in HbA1c levels.
ratio of patients who reached the HbA1c target of equal to or below 7% | Three months
  Comparison of the patient groups in their success in reaching the HbA1c target of equal to or below 7%.

SECONDARY OUTCOMES:
The effect of education on the HbA1c changes | Three months
  The effect of education on HbA1c changes and comparisons between the patient groups.
The effect of depression on the HbA1c changes | Three months
  The effect of depression as evaluated with Beck depression test on HbA1c changes and comparisons between the patient groups.
The effect of the level of physical activity on the HbA1c changes | Three months
  The effect of physical activity assessed by General practice physical activity questionnaire on HbA1c changes and comparisons between the patient groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse N Erbakan, MD, Principal Investigator — Istanbul Goztepe Prof. Dr. Suleyman Yalcin City Hospital
Locations (1):
- Istanbul Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Diabetes Association. 6. Glycemic Targets: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S73-S84. doi: 10.2337/dc21-S006. PMID 33298417
- [Background] Walraven I, Mast MR, Hoekstra T, Jansen AP, van der Heijden AA, Rauh SP, Rutters F, van 't Riet E, Elders PJ, Moll AC, Polak BC, Dekker JM, Nijpels G. Distinct HbA1c trajectories in a type 2 diabetes cohort. Acta Diabetol. 2015 Apr;52(2):267-75. doi: 10.1007/s00592-014-0633-8. Epub 2014 Oct 8. PMID 25287012
- [Background] Nichols GA, Joshua-Gotlib S, Parasuraman S. Glycemic control and risk of cardiovascular disease hospitalization and all-cause mortality. J Am Coll Cardiol. 2013 Jul 9;62(2):121-127. doi: 10.1016/j.jacc.2013.04.031. Epub 2013 May 9. PMID 23665365
- [Background] Satman I, Omer B, Tutuncu Y, Kalaca S, Gedik S, Dinccag N, Karsidag K, Genc S, Telci A, Canbaz B, Turker F, Yilmaz T, Cakir B, Tuomilehto J; TURDEP-II Study Group. Twelve-year trends in the prevalence and risk factors of diabetes and prediabetes in Turkish adults. Eur J Epidemiol. 2013 Feb;28(2):169-80. doi: 10.1007/s10654-013-9771-5. Epub 2013 Feb 14. PMID 23407904
- [Background] Satman I, Imamoglu S, Yilmaz C; ADMIRE Study Group. A patient-based study on the adherence of physicians to guidelines for the management of type 2 diabetes in Turkey. Diabetes Res Clin Pract. 2012 Oct;98(1):75-82. doi: 10.1016/j.diabres.2012.05.003. Epub 2012 May 29. PMID 22652276